CLINICAL TRIAL: NCT02598973
Title: Effect of Exercise on Recovery in Drug-Induced Parkinsonism and Parkinson Disease
Brief Title: Effect of Exercise in Parkinsonism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N2012-W
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parkinson's Disease; Drug-induced Parkinsonism
Keywords: Parkinson Disease; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Active Comparator): aerobic walking
  Interventions: Behavioral: Exercise
- No exercise (No Intervention): normal activity

INTERVENTIONS:
Behavioral: Exercise — Aerobic walking
  Arms: Exercise

SUMMARY:
Parkinson's disease (PD) is a common neurodegenerative disorder affecting approximately 80,000 Veterans, representing a priority area for VA research. Current medicines for PD only improve symptoms, treatments that slow disease progression are needed, and earlier diagnosis of PD may be the key to their development. PD symptoms can be mimicked by medicines (most commonly antipsychotic drugs that block dopamine), and some of these patients actually have underlying "prodromal" PD that was "unmasked" years before it would have caused symptoms. This problem is increasing as these medicines are now used for common conditions including post-traumatic stress disorder and depression. The investigators will identify prodromal PD in patients with drug-induced symptoms using brain scans. These patients will be enrolled in a randomized clinical trial of aerobic exercise which slows progression in animal models of PD and has other health benefits. The investigators will measure the effect of exercise on symptoms, disease progression (using brain scans) and markers of PD risk (using blood tests). These studies will improve early PD diagnosis and potentially identify a way to slow progression of PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is an incurable neurodegenerative disorder affecting approximately 1 million US adults and about 80,000 Veterans. PD causes significant morbidity due to motor and non-motor symptoms across its prolonged course with an annual economic burden of $14 billion in the US alone. Motor symptoms associated with loss of dopaminergic neurons in PD may be temporarily improved with dopamine replacing medicines, but disease-modifying therapies that delay or prevent neuronal loss are lacking and sorely needed. Exercise is promising as a disease-modifying therapy because it protects dopaminergic neurons in animal models of PD and has been associated with measures of neuroplasticity in PD patients. Unfortunately, more than half of dopaminergic neurons in the substantia nigra are lost before motor symptoms occur making it difficult to identify patients early enough to benefit from potentially disease-modifying therapies. Early "prodromal" PD can be identified using non-motor features including olfactory dysfunction and other biomarkers such as dopamine transporter (DaT) brain imaging abnormalities that are apparent years before motor symptoms. However, these strategies would be difficult and costly to implement on a population level without first identifying high-risk individuals for screening. Commonly prescribed dopamine blocking antipsychotic drugs cause debilitating PD-like motor dysfunction that is difficult to treat, and in some patients this finding may serve as a "stress test" for failing dopaminergic networks unmasking symptoms long before they would normally appear. Identifying prodromal PD among drug-induced parkinsonism patients offers a unique and unexplored opportunity for early intervention.

In the proposed studies, the investigators will employ a tiered screening strategy with inexpensive and non-invasive olfactory testing in drug-induced parkinsonism patients followed by DaT imaging in individuals with olfactory impairment to identify a cohort of patients with presumed prodromal PD. Subjects with presumed prodromal PD will then be randomized to a home-based exercise intervention ({5} times weekly aerobic walking confirmed by remote activity monitors) or no intervention. In this cohort, the investigators will assess: 1) Short-term symptomatic effects of exercise on motor function in drug-induced parkinsonism using standard clinical measures (Unified Parkinson's Disease Rating Scale) and quantitative gait assessments after 8 weeks of intervention; 2) a potential disease-modifying effect after 52 weeks of exercise by comparing the rate of change in quantitative DaT imaging; and 3) the mechanisms and biochemical correlates of exercise-induced changes using a panel of serum biomarkers implicated in exercise and/or PD risk including brain-derived neurotrophic factor, uric acid, and apolipoproteinA1. Differences in the rate of change between groups will be assessed using independent samples t-tests and linear mixed-effects models adjusting for age and gender. The investigators' preliminary data demonstrates a strong association between olfactory impairment and abnormal DaT imaging in drug-induced parkinsonism. Based on power calculations allowing for 20% dropout, the investigators will screen approximately 250 drug-induced parkinsonism subjects using olfactory testing, with the expectation that approximately 88 will have abnormal DaT imaging and agree to participate in the intervention trial.

Antipsychotic drugs are widely prescribed for a growing list of approved indications and off-label uses including bipolar disorder, depression and post-traumatic stress disorder. Studying drug-induced parkinsonism patients with prodromal PD will allow us to identify which individuals are at risk, characterize the natural history of progression and evaluate appropriate management strategies at the earliest stages of PD. Exercise as a putative disease-modifying therapy offers significant advantages including cost, ease of access and lack of toxicity compared with unproven pharmacologic interventions especially if offered early enough to have meaningful clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Subjects with parkinsonian signs:

  * rest tremor
  * rigidity
  * bradykinesia
* Parkinsonian signs occurring after the institution of therapy with a medication having a known association with DIP, examples include:

  * haloperidol
  * chlorpromazine
  * fluphenazine
  * perphenazine
  * risperidone
  * thioridazine
  * thiothixene
  * lithium
  * valproic acid
  * ziprasidone
  * olanzapine
  * aripiprazole
* Potential subjects with DIP will be pre-screened using a brief (12 item) scratch and sniff smell test with hyposmic subjects invited to learn more about the study.
* clinical diagnosis of H/Y <=2 PD

Exclusion Criteria:

* Subjects with a known diagnosis of atypical parkinsonian syndrome, i.e.:

  * dementia with Lewy bodies
  * progressive supranuclear palsy
  * corticobasal degeneration
  * multiple system atrophy)
  * or other neurodegenerative condition
* Subjects with a history of:

  * sinus trauma or surgery
  * encephalitis
  * current nasal congestion or other known reason for olfactory impairment
* Subjects with a contraindication to DaTI (sensitivity or allergy to iodine, treatment with a drug with a significant effect on DaTscan that cannot be temporarily weaned)
* Subjects with known unstable cardiac, pulmonary, orthopedic or other conditions that would preclude safe participation in exercise training
* Subjects currently engaging in exercise more than 45 minutes per day, 3 days per week

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Morley, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects underwent DAT-SPECT screening was part of the study protocol. Only subjects with positive DAT-SPECT were eligible to be randomized to one of the intervention arms. 9 were positive and started the exercise trial.
Period: Overall Study
Arm/Group | Exercise | No Exercise
Started | 5 (9 participants began the exercise phase) | 4
Completed | 3 | 3
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | No Exercise | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (6.8) | 61.5 (10.0) | 64.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Unified Parkinson's Disease Rating Scale Motor Exam [Mean (Standard Deviation); unit: units on a scale] — Standardized clinical exam scale. Minimum 0, Maximum 108. Higher scores indicate more severe Parkinson's symptoms.
  units on a scale | 17.3 (2.2) | 21.0 (5.4) | 19.3 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dopamine Transporter Imaging
Description: change in semi-quantitative Ioflupane-I123 uptake comparing exercise to no intervention.
Time Frame: 1 year
Population: Although 9 patients were enrolled in the exercise phase of the trial, only 6 (3 exercise arm, 3 control arm) completed the protocol and had a second imaging study to allow analysis of change over time
Measure: Mean (Standard Deviation); unit: % change in arbitrary intensity units
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 3 | 3
% change in arbitrary intensity units | 4.6 (22.0) | -15.9 (9.1)

2. Secondary Outcome: Change in Overall Motor Function
Description: change in UPRS motor exam at 8 weeks. Minimum 0, Maximum 108. Higher scores indicate more severe disease.
Time Frame: 8 weeks
Population: although 9 subjects enrolled, only 6 completed the protocol
Measure: Mean (Standard Deviation); unit: % change in score from baseline
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 3 | 3
% change in score from baseline | -2.3 (4.6) | 10.5 (10.6)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study entry until the end of study participation via weekly calls or spontaneous reporting over an average of 1 year
Description: per IRB definitions
Arm/Group | Exercise | No Exercise
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4
Other Adverse Events (participants affected / at risk) | 2/5 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=5) | No Exercise (N=4)
cancer diagnosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — subject was diagnosed with gastric cancer shortly after enrollment, before exercise testing
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=5) | No Exercise (N=4)
abnormal baseline exercise testing (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02598973/Prot_SAP_000.pdf